CLINICAL TRIAL: NCT03254329
Title: Establishing Global Reference Values for Human Milk Composition in a Multi-Center Collaborative Study
Brief Title: Establishing Global Reference Values for Human Milk
Acronym: MILQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of Copenhagen (Other); Medical Research Council Unit, The Gambia (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Universidade Federal do Rio de Janeiro (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MILQ
Record Dates: First submitted 2017-08-03; First posted 2017-08-18 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Human Milk Nutrient Reference Values
Keywords: human milk; micronutrients; lactation; milk volume; milk composition; reference values
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast milk, blood, saliva, urine and feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Bangladesh: Assessment of human milk nutrient composition. Approximately 500 women and their infants recruited, 250 dyads completing study
  Interventions: Other: Assessment of human milk nutrient composition
- Brazil: Assessment of human milk nutrient composition. Approximately 500 women and their infants recruited, 250 dyads completing study
  Interventions: Other: Assessment of human milk nutrient composition
- Denmark: Assessment of human milk nutrient composition. Approximately 500 women and their infants recruited, 250 dyads completing study
  Interventions: Other: Assessment of human milk nutrient composition
- The Gambia: Assessment of human milk nutrient composition. Approximately 500 women and their infants recruited, 250 dyads completing study
  Interventions: Other: Assessment of human milk nutrient composition

INTERVENTIONS:
Other: Assessment of human milk nutrient composition — Observational study to measure nutrients in human milk during lactation and their relationship to maternal and infant nutritional status.

SUMMARY:
The primary purpose of the proposed research is to establish Reference Values (RVs) for micronutrients (MN) and macronutrients in human milk. The investigators' research to date has revealed highly variable milk MN concentrations among populations, and very low values in some low income countries (LICs) likely caused by poor maternal status and/or diet but RVs are needed to interpret these values. During the past year the investigators conducted a review of human milk nutrient composition, and formed a Technical Advisory Group (TAG) which developed the current proposal. Here, the investigators are conducting a longitudinal project on well-nourished women and infants. The Mothers, Infants and Lactation Quality (MILQ) study is a multi-center cohort project, investigating breast milk nutrient composition in well-nourished women across the first 8.5 months of lactation in four different populations. The countries involved are Denmark, Brazil, Bangladesh and The Gambia. Exclusive breastfeeding is an eligibility criterion up until the second post-partum study visit (between 1 - 3.4 months postpartum), with the exception of the first week after delivery. Other data collected on mothers and infants, including maternal and infant nutrient intake and status, morbidity, milk volume, and infant development, will inform interpretation and support application of the results. While the priority is to develop RVs for MN, other analyses will include human milk oligosaccharides (HMOs) and proteins, and free amino acids (FAA) in infant plasma. Thus, with the samples obtained the investigators will perform (a) laboratory analyses of milk, plasma and urine nutrients to construct RVs for global application, (b) analyses of HMOs and proteins in milk, and (c) metabolomic analysis of FAA and other metabolites in infant plasma. By request of the Bill and Melinda Gates Foundation (BMGF), colostrum and fecal microbiota samples will also be collected and stored for later analyses.

DETAILED DESCRIPTION:
The investigators will collect breast milk samples at four visits, at 2-3 days after birth (colostrum) and at 1-3.4, 3.5-5.9, and 6-8.5 months of lactation from well-nourished mothers age ≥18 to ≤40 years, in a systematic, identical way in four countries. The four sites are: Copenhagen, Denmark; Banjul, The Gambia; Rio de Janeiro, Brazil; and Mirpur, Dhaka, Bangladesh. The most important site selection criteria were that multiple micronutrient supplements are not consumed after week 28 of pregnancy; maternal diet is adequate but consumption of highly fortified foods is limited; and exclusive breastfeeding is 60% at 4 months.

In order to have 250 women and infants per site complete the study at 8.5 months, approximately 500 women will be recruited during the third trimester of pregnancy. This should allow for mothers and infants not meeting study eligibility criteria in pregnancy or early lactation, and drop-outs from the study. Recruitment during pregnancy will increase the opportunity to locate and recruit women since recruitment in the immediate post-delivery period will be difficult. It will also enable the women to be counselled on the importance of exclusive breastfeeding (EBF). Colostrum will be collected at 2-3 days postpartum for future analysis. The first collection of mature milk will occur between 1 and 3.4 months postpartum, when maternal and infant blood samples will also be collected on all participants. At the final two visits, in addition to milk collection, blood will be taken from all mothers but only half of the infants each time, primarily for the assessment of micronutrient status.

A requirement is that infants must be EBF in the 1-3.4 month period, and breastfed (BF) in the second and third period. Longitudinal measurements on the same mother after the BF period are not necessary for statistical reasons, as the investigators are not creating RVs for change in milk composition. The investigators expect that due to attrition and cessation of BF, the sample size will need to be augmented in later months; the alternative would have been to recruit and measure many more women in earlier stages in order to have an adequate sample size in the 7-8.5 month interval, which would be a much less efficient approach. Therefore after 6 months, if women are not breastfeeding, additional lactating women will be recruited from the group that was not EBF in the 3.4 month period, or from the local health center or community.

At all three points of mature milk collection the investigators will measure breast milk volume; diet, anthropometry and morbidity of the mother and infant; and infant development at 3.5-5.9 and 6 to 8.5 months; and will collect infant fecal samples for future analyses of the microbiome. Milk volume will be measured at three sites using the International Atomic Energy Agency's protocol that requires dosing the mother with deuterated water and collecting maternal and infant saliva urine samples at 0, 1, 2, 3, 4, 13 and 14 days after the dose. In Denmark breast milk volume will be measured by 24 hour infant weighing.

Most of the laboratory analyses will be conducted at the United States Department of Agriculture, Agricultural Research Service, Western Human Nutrition Research Center (WHNRC) in Davis, California. Other analyses will be performed in the Department of Chemistry at University of California, Davis (HMOs and other bioactive compounds in milk), and the Swiss Federal Institute of Technology in Zurich (iodine status). RVs will be constructed following the methods and principles developed for the World Health Organization (WHO) Child Growth Standards and the Intergrowth-21st Project.

An add-on study "Evaluation of maternal insulin resistance, metabolic and inflammatory biomarkers for prediction of successful initiation and duration of breastfeeding" is being conducted at the Danish site and was approved by The Regional Committee on Health Research Ethics with (H-17015174).

The aims of the add-on study are to evaluate if maternal metabolic and inflammatory biomarkers can predict successful initiation and duration of breastfeeding in a population of healthy non-obese Danish women, to evaluate the impact of maternal inflammatory biomarkers during pregnancy on the offspring's growth and risk factors for later disease, and to relate the impact of maternal metabolic and inflammatory biomarkers during pregnancy on breastfeeding behavior and on the offspring's growth and risk factors for later disease in this population to corresponding outcomes in an established cohort of infants born of obese mothers.

ELIGIBILITY:
Inclusion Criteria for Mother

* No vitamin-mineral supplements during third trimester of pregnancy or during lactation except for iron + folic acid, also vitamin D and Ca in Denmark.
* Low habitual intake of highly-fortified foods (iodized salt excepted).
* No relevant past or current medical problems including gestational diabetes or pre-eclampsia.
* Singleton delivery, not preterm.
* BMI ≥18.5 to <30.0 kg/m2, height ≥150 cm.
* Mid-upper arm circumference (MUAC) ≥23 and ≤33 cm in pregnancy
* Consuming a nutritionally adequate diet i.e. not vegan or macrobiotic, ≥5 food groups/d each ≥15g. At screening this information will be collected with a locally-appropriate and validated food frequency questionnaire.
* Non-anemic in pregnancy (Hb >100 g/L)
* Alcohol intake ≤5 units (50 mL pure alcohol)/week.
* Non-smoker.

Inclusion Criteria for Infant

* Birth weight 2500-4200 g, 37-42 weeks of gestation.
* No congenital malformations that interfere with feeding or growth and development.

Exclusion Criteria at 1 to 3.4 Months Postpartum

* Cessation of or non-exclusive breastfeeding.
* Serious maternal illness.
* Infant length-for-age, weight-for-age or weight-for-length < -2 Z.

Exclusion criteria 3.5 to 8.5 months postpartum

* Cessation of breastfeeding.
* Serious maternal illness.
* Infant length-for-age, weight-for-age or weight-for-length < -2 Z.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant and lactating women
Study Population: Well-nourished pregnant women in the third trimester of pregnancy at recruitment, then lactating with their infant from 1-8.5 months postpartum.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in vitamin and mineral concentrations in human breast milk | Breast milk samples collected 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  To establish reference values, the vitamin and mineral concentrations will be measured in milk of well-nourished women

SECONDARY OUTCOMES:
Variation in other constituents of human breast milk | Breast milk samples collected at 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  Macronutrients, and human milk oligosaccharides and proteins will be analyzed
Micronutrient status of mothers and infants | Blood and urine samples surveyed at 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  Vitamin and mineral status of mothers and infants will be assessed in blood and urine
Milk volume | 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  Measurements of usual daily milk volume using deuterated water or, in Denmark, 24 hour infant weighing
Maternal and infant iodine status | 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  Urinary iodine; thyroid stimulating hormone, thyroglobulin and thyroxine in dried blood spots
Milk iodine | 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  Milk iodine
Maternal nutrient intake during pregnancy | Measured during gestational week 35-37
  Assessment of dietary intake by two days 24-hour recall in Denmark and Brazil
Maternal nutrient intake | 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  Assessment of dietary intake by two days 24-hour recall
Infant nutrient intake | 1-3.4, 3.5-5.9, and 6-8.5 months
  Assessment of dietary intake by two days 24-hour recall of the infant's diet
Infant dietary habits | 1-3.4, 3.5-5.9, and 6-8.5 months
  Assessment of dietary intake by diet habits questionnaire
Maternal weight | 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  Measure of weight in kilograms (kg)
Infant weight | 1-3.4, 3.5-5.9, and 6-8.5 months
  Measure of weight in grams (g) or kilograms (kg)
Maternal height | 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  measured in centimeters (cm)
Infant length | 1-3.4, 3.5-5.9, and 6-8.5 months
  measured in cm
Maternal body mass index | 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  Maternal weight and height will be combined to determine body mass index (kg/m2)
Infant growth | 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  Infant weight and length will be aggregated to determine infant growth status
Maternal body composition | 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  Assessment of body composition by bioimpedance in Denmark, The Gambia, and Brazil only.
Infant body composition | 1-3.4, 3.5-5.9, and 6-8.5 months
  Assessment of body composition by Air Displacement Plethysmography, in The Gambia, and by bioimpedance in Denmark and Brazil.
Infant morbidity | 1-3.4, 3.5-5.9, and 6-8.5 months
  Data collected from mothers on infant health
Infant development | 6-8.5 months
  Ages and Stages questionnaire
Infant motor development | 3.5-5.9 and 6-8.5 months
  Infant motor development measured using a World Health Organization (WHO) assessment of motor milestones
Change in infant microbiome | 1-3.4, 3.5-5.9, and 6-8.5 months
  DNA analyses of infant gut bacteria derived from fecal samples
Change in maternal microbiome | Collected at gestational week 28-40, and 1-3.4, 3.5-5.9, and 6-8.5 months postpartum
  DNA analyses of maternal gut bacteria derived from fecal samples in The Gambia and Brazil only
Maternal Glucose Tolerance | Measured once at gestational week 28-30
  In Denmark only, an Oral Glucose Tolerance Test will be performed. Fasting blood sugar (BS), and BS at 1 and 2 hours after glucose beverage.
Maternal Hemoglobin A1c (HbA1c) | Measured once at gestational week 28-30
  In Denmark only, maternal Hemoglobin A1c will be measured in whole blood
Maternal markers of insulin sensitivity | Measured once at gestational week 28-30
  In Denmark only, a serum sample will be collected and stored for measurement of insulin (mU/l), c-peptide (pmol/l), and leptin (ng/l)
Maternal lipid panel | Measured once at gestational week 28-30
  In Denmark only, a serum sample will be collected and stored for measurement of a lipid profile including Total Cholesterol, High Density Lipoprotein-cholesterol, Low Density Lipoprotein-cholesterol, Very Low Density Lipoprotein-cholesterol, and Triglycerides in mmol/l).
Maternal inflammatory markers | Measured once at gestational week 28-30
  In Denmark only, a serum sample will be collected and stored for measurement of high sensitivity C-reactive protein (mg/l).

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay H Allen, PhD, Principal Investigator — USDA/WHNRC
Locations (4):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh
- Federal University of Rio de Janeiro, Rio de Janeiro, Brazil
- University of Copenhagen, Copenhagen, Frederiksberg, Denmark
- Medical Research Council Gambia, Bakau, Kombo Saint Mary's, The Gambia

IPD SHARING:
Plan to Share IPD: No
Individual participants data will only be available as de-identified data.

REFERENCES:
- [Derived] Christensen SH, Rom AL, Greve T, Lewis JI, Frokiaer H, Allen LH, Molgaard C, Renault KM, Michaelsen KF. Maternal inflammatory, lipid and metabolic markers and associations with birth and breastfeeding outcomes. Front Nutr. 2023 Sep 4;10:1223753. doi: 10.3389/fnut.2023.1223753. eCollection 2023. PMID 37731394
- [Derived] Christensen SH, Lewis JI, Larnkjaer A, Frokiaer H, Allen LH, Molgaard C, Michaelsen KF. Associations between maternal adiposity and appetite-regulating hormones in human milk are mediated through maternal circulating concentrations and might affect infant outcomes. Front Nutr. 2022 Nov 4;9:1025439. doi: 10.3389/fnut.2022.1025439. eCollection 2022. PMID 36407523
- [Derived] Allen LH, Hampel D, Shahab-Ferdows S, Andersson M, Barros E, Doel AM, Eriksen KG, Christensen SH, Islam M, Kac G, Keya FK, Michaelsen KF, de Barros Mucci D, Njie F, Peerson JM, Moore SE. The Mothers, Infants, and Lactation Quality (MILQ) Study: A Multi-Center Collaboration. Curr Dev Nutr. 2021 Sep 20;5(10):nzab116. doi: 10.1093/cdn/nzab116. eCollection 2021 Oct. PMID 34712893